CLINICAL TRIAL: NCT02073175
Title: Development of Dietary Supplements for Mood Symptoms in Postpartum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Program Head, Neurochemical Imaging for Mood Disorders, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112/2013
Record Dates: First submitted 2014-02-21; First posted 2014-02-27 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Postpartum Blues; Healthy
Keywords: Postpartum; Dietary Supplements; Mood Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Postpartum with crying spells-Full dose (Experimental): Healthy women who are within the first 18 months postpartum and have crying spells but do not have major depression. The effect of the dietary supplement in reducing sadness in this group will be assessed.
  Intervention: Full dose dietary supplement Motherwell
  Interventions: Drug: Motherwell
- Day-5 postpartum - Full dose (Experimental): Healthy women on day-5 postpartum. This group is recruited during pregnancy but the main study day, involving the dietary supplement consumption is being done after delivery and during postpartum.
  Intervention: Full dose dietary supplement Motherwell
  Interventions: Drug: Motherwell
- Day-5 postpartum - Half dose (Experimental): Healthy women on day-5 postpartum. This group is recruited during pregnancy but the main study day, involving the proposed dietary supplement consumption, is being done after delivery and during postpartum.
  Intervention: Half dose dietary supplement Motherwell
  Interventions: Drug: Motherwell
- Day-5 postpartum - Quarter dose (Experimental): Healthy women on day-5 postpartum. This group is recruited during pregnancy but the main study day, involving the proposed dietary supplement consumption, is being done after delivery and during postpartum.
  Intervention: Quarter dose dietary supplement Motherwell
  Interventions: Drug: Motherwell
- Day-5 postpartum - Control (Other): Healthy women on day-5 postpartum. This group is recruited during pregnancy but the main study day, involving a control supplement consumption, is being done after delivery and during postpartum.
  Intervention: Control protein to compare with Motherwell
  Interventions: Drug: Motherwell

INTERVENTIONS:
Drug: Motherwell — The interventions involves a dietary supplement called Motherwell, at current stage, to reduce the intensity of sadness in women vulnerable to sadness.

SUMMARY:
The purpose of this study is to determine whether a dietary supplement (DS) is effective in protecting against sad mood in postpartum.

DETAILED DESCRIPTION:
The specific aim of this open-label study is to assess whether the proposed dietary supplement can reduce the intensity of sadness in women vulnerable to sadness (day-5 postpartum women and women within the first 18 months postpartum with crying spells).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45
* The subject, as reported by them, should be in a good health.
* The subject is not taking any medication.
* The subject is not taking any investigational medicinal product within 8 weeks.
* BMI 19 to 40 (kg/m2)
* Resting pulse between 45 and 100 bpm
* Systolic blood pressure between 91 and 139 mmHg (inclusive)
* Diastolic blood pressure between 51 and 90 mmHg (inclusive)

Exclusion Criteria:

* The subject has been diagnosed with any axis 1 and 2 disorders based on Structured Clinical Interview (SCID) for DSM-IV interview.
* Substance abuse disorder
* Subjects who have been smoking in the past 5 years.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) | Assessment will be done on day-5 postpartum or within the first 18 months postpartum (depending on which group subject belongs to). On the assessment day, the VAS will be administered before and after sad mood indcution and compared
  VAS uses a 10-cm scale for participants to indicate the extent to which each of them feel happy or sad. The change in VAS before versus after sad mood induction is the change score in VAS. The change score on the day with active dietary supplement is compare to the change score of the subjects who have not received any supplement and have been recently recruited

SECONDARY OUTCOMES:
Change in Profile of Mood States (POMS) Scores | Assessment will be done on day-5 postpartum or within the first 18 months postpartum (depending on which group subject belongs to). On the assessment day, the POMS will be administered before and after sad mood indcution and compared
  The POMS contains 65 adjectives rated by participants on a 5-point scale. Six factors are derived that include tension, depression, anger, fatigue, vigor and confusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Meyer, MD,PhD,FRCPC, Principal Investigator — Research Imaging Centre, Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiciton and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowlati Y, Ravindran AV, Segal ZV, Stewart DE, Steiner M, Meyer JH. Selective dietary supplementation in early postpartum is associated with high resilience against depressed mood. Proc Natl Acad Sci U S A. 2017 Mar 28;114(13):3509-3514. doi: 10.1073/pnas.1611965114. Epub 2017 Mar 13. PMID 28289215
- See also: Information about research at the Centre for Addiction and Mental Health — http://camh.ca/research